CLINICAL TRIAL: NCT00994877
Title: Thromboelastography in Patients Admitted to the ICU for Severe Sepsis
Brief Title: Thromboelastography in in Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: ASAF MILLER MD, Assaf Harofeh Medical Center
Other Study IDs: 34/09
Record Dates: First submitted 2009-09-24; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Shock, Surgical; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Shock, Surgical; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Septic Patients
- Healthy Control

SUMMARY:
Methods:

The study is an observational prospective trial that includes 150 patients 18 or older admitted to our icu because of severe sepsis or septic shock as defined by the American College of Chest Physicians/ Society of Critical Care Medicine consensus conference.

Patients whose primary reason for hospital admission is sepsis or patients developing sepsis after elective invasive procedure will be included.

Only patients with known former primary coagulation/hypercoagulability disorder wil be excluded.

Procedure:

Within 12 hours of admission to the intensive care unit (ICU) blood will be drawn for the following:

Blood count, glucose, urea, creatinine, liver function tests, prothrombin time, partial thromboplastin time, Ddimer, fibrinogen and TEG (thromboelastography) assay will be performed.

These blood tests will be also drawn on day 2 and 4 of admission. On day one, another 3 cc of blood will be drawn and frozen in -80 degrees for levels of coagulation factors: I, II, V, VII, VIII, IX, X, XI, XII, XIII, Antithrombin III, protein C, S.

Demographic data will be collected according to patient chart, and the acute physiologic and chronic health evaluation (APACHE) II score will be assessed after 24 hours. Vital signs will be collected from monitors.

Informed consent will be waved due to lack of any intervention and the general condition of patients unable to sign an informed consent.

Control group will include 10 healthy individuals.

End point:

The primary end point is to determine the common hypercoagulable/coagulation disorders according to TEG.

The secondary end point is to determine whether TEG results have prognostic implications on this group of severe septic patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 years or older admitted to ICU whose primary reason for admission was sepsis or suffering sepsis or septic shock after elective surgical procedure

Exclusion Criteria:

* Patients suffering primary disease affecting the coagulation system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients With sepsis or septic shock admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
To determine the common hypercoagulable/ coagulation disorders according to thromboelastography (TEG) | In hospital

SECONDARY OUTCOMES:
To determine whether TEG results have prognostic implications on this group of severe septic patients | 28 day

CONTACTS AND LOCATIONS:
Overall Officials: asaf miller, md, Principal Investigator — Asaf Harofeh Medical Center
Locations (1):
- Asaf Harofeh Medical Center, Beer Yaakov, Israel

REFERENCES:
- [Background] Martini WZ, Cortez DS, Dubick MA, Park MS, Holcomb JB. Thrombelastography is better than PT, aPTT, and activated clotting time in detecting clinically relevant clotting abnormalities after hypothermia, hemorrhagic shock and resuscitation in pigs. J Trauma. 2008 Sep;65(3):535-43. doi: 10.1097/TA.0b013e31818379a6. PMID 18784565